CLINICAL TRIAL: NCT04828746
Title: Utility of Ultrasound-Guided Site Marking in Pediatric Lumbar Punctures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carilion Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB-20-800
Record Dates: First submitted 2021-03-26; First posted 2021-04-02 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Ultrasound Therapy; Complications

STUDY DESIGN:
Intervention Model Description: Patients assigned to either pre-procedural ultrasound-guided anatomy review and skin marking prior to a lumbar puncture v standard of care, palpation only guided lumbar puncture.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients who will undergo lumbar puncture without pre-procedural ultrasound-guided skin marking
- Experimental (Experimental): Patients who will undergo lumbar puncture after pre-procedural ultrasound-guided skin marking
  Interventions: Procedure: Ultrasound Guided Skin Marking

INTERVENTIONS:
Procedure: Ultrasound Guided Skin Marking — Using ultrasound for skin marking pre-procedure
  Arms: Experimental

SUMMARY:
The standard way to identify landmarks in the spine before inserting a needle for a lumbar puncture is to feel by touch. The purpose of this research is to determine if doing an ultrasound to identify landmarks before performing a lumbar puncture will improve the first-time success rate of the needle insertion in pediatric patients.

DETAILED DESCRIPTION:
Subjects will be identified for the study after meeting inclusion & exclusion criteria. Part of said criteria is that the patient will medically require a lumbar puncture (LP) to be completed for their medical care and the patient is currently located in the Carilion Roanoke Memorial Hospital (CRMH) Pediatric Emergency Department, Pediatric Ward, or Pediatric Intensive Care Unit. After the study team member identifies a patient who meets the criteria and obtains the necessary consent/assent(s) the practitioner will then load the preset procedure note into the electronic medical record. In this procedure note, there will be a link to REDCap (a secure data collection tool) where the study team member will enter the patient's medical record number and date of birth. The participant will then be randomized to either the standard of care/ control group (palpation only lumbar puncture) or the experimental group (lumbar puncture after ultrasound-guided (US) skin marking) via REDCap. REDCap will be set to randomize participants via block randomization to the desired total number of 60 (30 in each control and experiential groups), and no study team member/ practitioner will have access to the set block randomization parameters in REDCap.

Regarding sedation versus analgesia (performed for standard of care reasons and not affected by the research study), the decision on what is best and needed for the patients will be up to the performing practitioner in both groups. This ranges from superficial skin numbing cream and sucrose gel (for neonates) to lidocaine injections to oral or IV medications for pain/anxiety to full procedural sedation; or a combination of any of these methods. This will be entirely up to the performing practitioner as the methods used can vary greatly from patient to patient based on a multitude of factors. If procedural sedation is required then often another attending physician must be present in order to administer the sedating medications but this individual is not part of the study and will obtain their own consent for sedation as applicable as per Carilion Clinic policy. The agent(s) of choice will be clearly documented in the procedure note so this information can be taken into consideration when performing data analysis. All sedation v analgesia will take place prior to beginning the procedure. Once the practitioner is ready to begin they will start a timer to properly keep time as to the duration of the entire procedure.

The practitioner performing the lumbar puncture procedure will either be a study team member or another practitioner who is under the direct supervision of a study team member (e.g. advanced care practitioner under an attending, a junior resident under a senior resident). The study team member will supervise/perform the procedure as indicated to not only ensure the safety of patients but to make sure proper protocol is followed.

After analgesia v sedation is administered, if the participant is in the standard of care group, the practitioner will then position the patient in the best position they believe is needed to obtain the cerebral spinal fluid (CSF) sample. This is typically sitting upright or having the patient lying down on their side (with the latter being more common). The practitioner will then palpate the area they feel is the best to insert the spinal needle to collect the sample. The gap that is being palpated is typically between the 3rd and 4th or the 4th and 5th lumbar vertebrae. Following this, the practitioner will then don sterile gloves, and clean the patient's back with betadine or chlorhexidine as per their discretion. The spinal needle will then be inserted into the spinal interspace, the stylet from the needle will be removed, and the fluid will be collected. The amount of fluid that will be collected varies based on the patient's age as well as the testing that is deemed clinically necessary. Typically 1-3 milliliters of CSF will be collected in each of the 3-4 tubes that are provided in the LP kit that is used for the procedure. After the fluid is collected, the needle will then be removed and pressure will be held on the insertion site to ensure no bleeding or CSF leakage. When bleeding or fluid leakage has halted the procedure is then completed and the timer is stopped. The time it takes to perform this procedure varies greatly with different practitioners and patients but is typically completed within 15-60 minutes.

After analgesia v sedation is administered, if the participant is in the experimental group (use of ultrasound), the practitioner will then position the patient in the best position they believe is needed to obtain the cerebral spinal fluid (CSF) sample. This is typically sitting upright or having the patient lying down on their side (with the latter being more common). The practitioner will then use a portable, point-of-care US machine in order to identify the best interspace to obtain the sample. This involves using a small amount of US gel (a non-toxic, water-based substance used to improve sound waves and therefore picture quality when performing the US) and the actual US probe on the patient's back. After the desired space is identified in the sagittal and transverse planes with the US machine, a small mark will be placed on the patient using a surgical pen (a marker similar to a "sharpie" but is safe for use on human skin and will wash off in 1-2 days). The desired space that is being identified is typically between the 3rd and 4th or the 4th and 5th lumbar vertebrae. Following this, the practitioner will then wipe the US gel off the patient's back, don sterile gloves, and clean the patient's back with betadine or chlorhexidine as per their discretion. The spinal needle will then be inserted into the spinal interspace that was identified and marked as noted previously, the stylet from the needle will be removed, and the fluid will be collected. The amount of fluid that will be collected varies based on the patient's age as well as the testing that is deemed clinically necessary. Typically 1-3 milliliters of CSF will be collected in each of the 3-4 tubes that are provided in the LP kit that is used for the procedure. After the fluid is collected, the needle will then be removed and pressure will be held on the insertion site to ensure no bleeding or CSF leakage. When bleeding or fluid leakage has halted the procedure is then completed and the timer is stopped. The time it takes to perform this procedure varies greatly with different practitioners and patients but we anticipate it taking between 25-70 minutes. The extra time allotted is due to the use of the US, but how much time exactly it will take is not fully known, and in fact, it may not add time as compared to the control population but this will need to be investigated further during data analysis. There is potential for a patient to be under sedation (as discussed above) for a longer time if using US rather than the standard of care palpation only, but this is currently unknown.

CSF will be sent to the lab and analyzed with the tests that are deemed needed by the practitioner. In general, it is commonplace for a "CSF Cell Count & Differential" to be ordered on all CSF samples as this is a baseline test of the sample. The data provided from this test will be analyzed by research team members via the medical record but the actual sample itself or what additional tests are ordered will in no way be impacted by the research. Specifically, this test tells the study team member how many red blood cells are present in the CSF. With some exceptions, the fewer red blood cells that are present in the CSF fluid is indicative of a procedure that was able to be performed smoothly, efficiently, and without multiple attempts. The CSF from the first tube will be used for the "CSF Cell Count & Differential", which again is commonplace. In some, uncommon instances (for various reasons including dehydration, failed LP attempt) only a small amount of CSF can be obtained. Should this be the case, the practitioner will decide what tests are needed on the small CSF sample. Data from the procedure (excluding the "CSF Cell Count & Differential" if there was not enough sample to run this test) may still be used in data analysis so the participant will still be enrolled in the study. An instance in which this may occur is on a dehydrated child where there are suspicions of meningitis. In this case, the most crucial test to run on the CSF is a bacteria or viral culture. Again the cell count and differential are still very helpful and standard to order on these samples but the first priority goes to the culture if there was only a small sample that was able to be obtained.

The amount of time needed to access the patient's medical record by a study team member after the procedure and lab test completion is approximately 30 minutes per patient. In general, the patient's age, weight, height, the results of the "CSF Cell Count & Differential" lab testing, the level of the practitioner but not their identity (ie resident v attending), and procedure notes will be specifically accessed for collection and analyzing. This will be done in a HIPAA compliant manner (e.g. private, secure, password-protected computers, internet access, and databases). At least weekly a member of the study team will be accessing patient charts (with the HIPAA data provided by REDCap) in order to extract the de-identified data required and place it in a secure spreadsheet. After the de-identified data is collected, the participant's medical chart, as well as PHI, will not need to be accessed again. No follow-up will be needed for the purposes of this study.

ELIGIBILITY:
Inclusion Criteria:

* Birth to 17y of age
* Patient currently in Pediatric ED, Ward, or ICU
* Determined by providers caring for the patient that lumbar puncture is clinically indicated
* Parent/Legal Guardian able to give consent prior to the procedure

Exclusion Criteria:

* Known anatomic spinal deformity (e.g. scoliosis)
* Critical illness where emergent lumbar puncture is needed
* Patients only able to be entered in the study once per encounter
* Patients who are wards of the state or in foster care

Max Age: 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Attempts | Through study completion, anticipated average of 1 year
  Number of attempts required for successful LP and subsequent specimen collection

SECONDARY OUTCOMES:
Age | Through study completion, anticipated average of 1 year
  Documented age 0-17 years
BMI | Through study completion, anticipated average of 1 year
  Evaluate BMI v success rate
LP Position | Through study completion, anticipated average of 1 year
  Evaluate position for lumbar puncture
Quality of CSF sample based on grading criteria | Through study completion, anticipated average of 1 year
  Grade of CSF Sample Criteria for Grading
  Grade I
  <250 Red Blood Cells (RBCs)
  Grade II
  250-1000 RBCs
  Grade III
  1000-5000 RBCs
  Grade IV
  >5000 RBCs
Time required for procedure completion | Through study completion, anticipated average of 1 year
  Evaluate if adding ultrasound increases time of procedure in total

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Pandey, MD, Principal Investigator — Carilion Clinic Physician
Locations (1):
- Carilion Roanoke Memorial Hospital, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No